CLINICAL TRIAL: NCT02147353
Title: An Investigator-Initiated Study to Assess the Safety and Efficacy of Sinecatechins 15% Ointment When Used in Conjunction With Cryotherapy in the Treatment of External Genital Warts
Brief Title: Treatment of External Genital Warts With Cryotherapy and Sinecatechins 15% Ointment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Principal Investigator, Gary Goldenberg, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 11-0860
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: External Genital Warts
Keywords: External Genital Warts; Sinecatechins; Cryotherapy
MeSH Terms: interventions — green tea extract polyphenone E; Ointments; Cryotherapy; Cryosurgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sinecatechins 15% Ointment & Cryotherapy (Active Comparator): Cryotherapy and then Sinecatechins 15% Ointment 1 week later.
  Interventions: Drug: Sinecatechins 15% Ointment; Drug: Cryotherapy alone
- Cryotherapy Alone (Placebo Comparator): Cryotherapy will be standardized in all subjects and for all treated lesions: EGW lesions will be treated with 2 sprays, 5 seconds each, with a 5 second interval. All subjects will be treated with the same cryo-spray regimen.
  Interventions: Drug: Cryotherapy alone

INTERVENTIONS:
Drug: Sinecatechins 15% Ointment — Following cryotherapy, half of the subjects will be randomized to treatment with sinecatechins ointment twice daily starting one week after cryotherapy (Week 1).
  Other Names: Veregen
  Arms: Sinecatechins 15% Ointment & Cryotherapy
Drug: Cryotherapy alone — Cryotherapy will be standardized in all subjects and for all treated lesions.
  Other Names: Cryosurgery

SUMMARY:
External Genital Warts (EGW) are the most common sexually transmitted disease associated with more than 30 types of the Human Papillomavirus (HPV). Cryotherapy is an effective method of EGW treatment. However, multiple sessions may be required with reported clearance rates ranging between 27-88%. Sinecatechins 15% ointment is Food and Drug Administration approved for three times daily application in immunocompetent subjects 18 years and older for the treatment of EGW and perianal warts. Treatment of EGW with cryotherapy followed by sinecatechins appears to be logical. Cryotherapy has direct cytodestructive effects with immediate short-term efficacy on treated EGW, while sinecatechins provide field therapy, treating both clinical and sub-clinical lesions. For this study, the investigators used sinecatechins 15% ointment twice daily regimen and anticipated that the synergistic effect with cryotherapy will provide better efficacy that cryotherapy alone. The investigators also anticipated that the sequential therapy with be safe.

DETAILED DESCRIPTION:
A total of 42 subjects received standardized cryotherapy to all lesions, using two cycles of five seconds each, separated by a five second interval rest (Week 0/Baseline). One week following cryotherapy, subjects were randomized 1:1 to either additional treatment with sinecatechins 15% ointment twice daily or no additional treatment. Those subjects randomized to additional treatment received sinecatechins 15% ointment BID for up to sixteen weeks, or until complete clearance of all EGW, whichever occurred first. Additionally, subjects were advised to maintain safe sexual practices and have all recent sexual partners examined for EGW. Subjects were followed every 8 weeks for a total of 16 weeks (Table 1). EGW lesion counts were conducted at all study visits by the same qualified blinded evaluator. Additionally, at each visit local skin reactions, change in concomitant medications, and adverse events were assessed. Any subjects who received sinecatechins 15% ointment and discontinued prematurely were asked to return for an End of Study Visit. Females of childbearing potential underwent a urine pregnant test at all visits during study treatment period. Subjects that met complete responder criteria as above, were additionally followed and assessed at Visit5/Week 41 and Visit 6/Week 65 to assess for wart recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years old with at least two visible EGWs.
* Subject must be in good general health as confirmed by the medical history.
* Subject must be able to read, sign, and understand the informed consent.
* Subject must be willing to forego any other treatments for his/her EGW lesions.
* Subject is willing and able to participate in the study as an outpatient, making frequent visits to the study center during the treatment and follow-up periods and to comply with all study requirements including concomitant medication and other treatment restrictions.
* If subject is a female of childbearing potential she must have a negative urine pregnancy test result prior to study treatment initiation and must agree to use an approved method of birth control while enrolled in the study.

Exclusion Criteria:

* Subject with any evidence of herpes genitalis or any other current and/or recurrent genital or uncontrolled infection, including Human Immunodeficiency Virus, Hepatitis B or Hepatitis C.
* Subject with an unstable medical condition as deemed by the clinical investigator.
* Subject with any dermatologic disease in the treatment area that may be exacerbated by the treatment proposed or that might impair the evaluation of EGW lesions.
* Subject who has previously been treated in an EGW clinical trial, had treatment of anogenital warts or had systemic intake of virostatics or immunosuppressive medication within 30 days prior to Baseline Visit.
* Women who are pregnant, lactating, or planning to become pregnant during the study period.
* Subject who have experienced a clinically important medical event within 90 days of the visit (e.g., stroke, myocardial infarction, etc).
* Subject who have active chemical dependency or alcoholism as assessed by the investigator.
* Subject who have known allergies to any component of the study ointment.
* Subject who have organ allograft, skin conditions that may interfere with study ointment, or having internal (vaginal or rectal) warts that have required treatment.
* Subject who has received any of the following within 90 days prior to study treatment initiation:

  * interferon or interferon inducers
  * cytotoxic drugs
  * immunomodulators or immunosuppressive therapies (inhaled/ intranasal corticosteroids are permitted)
  * oral or parenteral corticosteroids
  * topical corticosteroids if greater than 2 gm/day
  * any dermatologic procedures or surgeries on the study area (including any EGW treatments)
* Subject who have used any topical prescription medications on the study area within 30 days prior to study treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Goldenberg, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] On SC, Linkner RV, Haddican M, Yaroshinsky A, Gagliotti M, Singer G, Goldenberg G. A single-blinded randomized controlled study to assess the efficacy of twice daily application of sinecatechins 15% ointment when used sequentially with cryotherapy in the treatment of external genital warts. J Drugs Dermatol. 2014 Nov;13(11):1400-5. PMID 25607709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were enrolled from September 2011 to December 2012.
Groups:
- Sinecatechins 15% Ointment & Cryotherapy: Cryotherapy and then Sinecatechins 15% Ointment 1 week later.
  Sinecatechins 15% Ointment: Following cryotherapy, half of the subjects randomized to treatment with sinecatechins ointment twice daily starting one week after cryotherapy up to 16 weeks or until complete clearance.
- Cryotherapy Alone: Cryotherapy standardized in all subjects and for all treated lesions: EGW lesions treated with 2 cycles, 5 seconds each, with a 5 second interval. All subjects treated with the same cryo-spray regimen.
Period: Overall Study
Arm/Group | Sinecatechins 15% Ointment & Cryotherapy | Cryotherapy Alone
Started | 21 | 21
Completed | 12 | 21
Not Completed | 9 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — unable to make visits | 4 | 0
Not completed — medication noncompliance | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sinecatechins 15% Ointment and Cryotherapy: Sinecatechins 15% Ointment: Following cryotherapy, half of the subjects randomized to treatment with sinecatechins ointment twice daily starting one week after cryotherapy up to 16 weeks or until complete clearance.
- Total: Total of all reporting groups
Arm/Group | Sinecatechins 15% Ointment and Cryotherapy | Cryotherapy Alone | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (5.2) | 35.8 (4.4) | 37.3 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Clearance,
Description: Subjects with complete clearance, or no longer have HPV infected cells. Complete clearance was defined as zero lesions at the respective time points.
Time Frame: at week 1, week 9, and week 17
Measure: Number; unit: participants
Arm/Group | Sinecatechins 15% Ointment & Cryotherapy | Cryotherapy Alone
Number analyzed (Participants) | 21 | 21
participants
  at week 1 | 0 | 0
  at week 9 | 3 | 5
  at week 17 | 6 | 6

2. Secondary Outcome: Number of Participants With Recurrence of Previously Treated EGW Lesions
Description: To evaluate the efficacy of using combination cryotherapy-sinecatechins 15% ointment BID versus cryotherapy alone on EGW lesions via recurrence rates of previously treated EGW lesions in those subjects who achieved a complete response over a 24 week post-treatment period.
Time Frame: at 24 week post-treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Sinecatechins 15% Ointment & Cryotherapy | Cryotherapy Alone
Number analyzed (Participants) | 21 | 21
Participants | 1 | 5

3. Secondary Outcome: Number of Participants With Recurrence of Previously Treated EGW Lesions
Description: To evaluate the efficacy of using combination cryotherapy-sinecatechins 15% ointment BID versus cryotherapy alone on EGW lesions via recurrence rates of previously treated EGW lesions in those subjects who achieved a complete response over a 48 week post-treatment period.
Time Frame: at 48 week post-treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Sinecatechins 15% Ointment & Cryotherapy | Cryotherapy Alone
Number analyzed (Participants) | 21 | 21
Participants | 2 | 6

4. Secondary Outcome: Local Skin Reactions
Description: To evaluate the safety of cryotherapy-sinecatechins 15% ointment BID versus cryotherapy alone as a regimen for EGW by evaluating for local skin reactions and adverse events.
  Number of participants with local skin reactions.
Time Frame: at 16 week treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Sinecatechins 15% Ointment & Cryotherapy | Cryotherapy Alone
Number analyzed (Participants) | 21 | 21
Participants | 21 | 21

5. Secondary Outcome: Subjects With Partial Clearance of Lesions
Description: Partial clearance is described as at least 50% reduction from baseline
Time Frame: At week 1, week 9, and week 17
Measure: Number; unit: participants
Arm/Group | Sinecatechins 15% Ointment & Cryotherapy | Cryotherapy Alone
Number analyzed (Participants) | 21 | 21
participants
  at week 1 | 7 | 6
  at week 9 | 15 | 9
  at week 17 | 15 | 11

6. Secondary Outcome: Mean Change in Number of Lesions
Description: Mean change in number of lesions after 1 weeks, 9 weeks and 17 weeks post treatment as compared to baseline
Time Frame: Week 1, week 9 and week 17
Population: data for only those participants who returned for the respective visits.
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Sinecatechins 15% Ointment & Cryotherapy | Cryotherapy Alone
Number analyzed (Participants) | 21 | 21
number of lesions
  Week 1 | -2.2 (3.93) | -2.1 (3.83)
  Week 9: number analyzed (Participants) | 20 | 18
  Week 9 | -5.4 (5.71) | -2.7 (3.68)
  Week 17: number analyzed (Participants) | 15 | 10
  Week 17 | -4.8 (7.87) | -3.8 (5.49)

7. Secondary Outcome: Mean Change in Number of Lesions
Description: Mean change in number of lesions as compared to baseline at Week 1, Week 9 and Week 17 for the intent-to-treat population
Time Frame: At week 1, week 9, and week 17
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Sinecatechins 15% Ointment & Cryotherapy | Cryotherapy Alone
Number analyzed (Participants) | 21 | 21
lesions
  Week 1 | -2.2 (3.93) | -2.1 (3.83)
  Week 9 | -5.0 (5.74) | -2.1 (3.75)
  Week 17 | -5.0 (6.90) | -2.1 (4.73)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 65 weeks
Description: There were no serious adverse events related to the study medication reported during the study. All subjects experienced mild to moderate local site reactions (eg, any symptom of erythema, edema, scaling, crusting, and erosion which were not collected separately) that were related to both cryotherapy and/or sinecatechins ointment. There were no subject discontinuations or dose interruptions.
Arm/Group | Sinecatechins 15% Ointment & Cryotherapy | Cryotherapy Alone
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 21/21 | 21/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sinecatechins 15% Ointment & Cryotherapy (N=21) | Cryotherapy Alone (N=21)
local site reactions (Skin and subcutaneous tissue disorders) | 21 (21) | 21 (21) — Local site reactions is any experienced mild to moderate local site reactions (erythema, edema, scaling, crusting, and erosion). these were not separated out.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes